CLINICAL TRIAL: NCT02703272
Title: A Randomized, Open-label, Safety and Efficacy Study of Ibrutinib in Pediatric and Young Adult Patients With Relapsed or Refractory Mature B-cell Non-Hodgkin Lymphoma
Brief Title: A Safety and Efficacy Study of Ibrutinib in Pediatric and Young Adult Participants With Relapsed or Refractory Mature B-cell Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: IDMC recommended that enrolment be stoped, as the EFS hazard ratio and associated p-value crossed the futility boundary specified in protocol (July 2020).
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108134; 54179060LYM3003 (Other: Janssen Research & Development, LLC); 2016-000259-28 (EudraCT Number)
Record Dates: First submitted 2016-03-03; First posted 2016-03-09 (Estimated); Results first posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Lymphoma, Non-Hodgkin; Ibrutinib; JNJ-54179060
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — ibrutinib; Rituximab; Ifosfamide; Carboplatin; Etoposide; Vincristine; Idarubicin; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Ibrutinib (Experimental): The first 2 participants enrolled in each age group (1-5 years, 6-11 years and 12-17 years) will receive starting dose of Ibrutinib 240 milligram per square meter (mg/m^2) for the first cycle, followed by dose escalation at the start of Cycle 2 as long as all pharmacokinetic assessments are within the expected range and there are no safety concerns. For participants being treated at 240 mg/m^2 dose level during the first cycle, the maximum dose should not exceed a total of 420 mg/day. All participants will receive rituximab, ifosfamide, carboplatin, etoposide and dexamethasone (RICE) or ituximab, vincristine, ifosfamide, carboplatin, idarubicin and dexamethasone (RVICI) background therapy (investigator's choice), during treatment phase. Participants with PR or better only will receive Ibrutinib for 3 cycles or until PD, unacceptable toxicity or until initiating antilymphoma therapy or a conditioning regimen for stem cell transplantation during post-treatment phase.
  Interventions: Drug: Ibrutinib; Drug: Rituximab; Drug: Ifosfamide; Drug: Carboplatin; Drug: Etoposide; Drug: Vincristine; Drug: Idarubicin; Drug: Dexamethasone
- Part 2: Ibrutinib (Experimental): Participants will either receive ibrutinib and RICE/RVICI background therapy or RICE/RVICI background therapy alone, until 3 cycles are completed or until PD or unacceptable toxicity during the treatment phase. Participants who received ibrutinib and RICE/RVICI background therapy and with PR or better only will receive ibrutinib alone for 3 cycles during post-treatment phase.
  Interventions: Drug: Ibrutinib; Drug: Rituximab; Drug: Ifosfamide; Drug: Carboplatin; Drug: Etoposide; Drug: Vincristine; Drug: Idarubicin; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ibrutinib — Participants will receive Ibrutinib (dose 240 mg/m^2 /329 mg/m^2 per day) during part 1 and part 2.
Drug: Rituximab — Participants will receive a cumulative dose of rituximab 750 mg/m^2 as a part of RICE/RVICI regimen in part 1 and part 2 per cycle.
Drug: Ifosfamide — Participants will receive a cumulative dose of Ifosfamide 9 g/m^2 and 10 g/m^2 as a part of RICE and RVICI regimen respectively in part 1 and part 2 per cycle.
Drug: Carboplatin — Participants will receive a cumulative dose of carboplatin 635 mg/m^2 and 800 mg/m^2 as a part of RICE and RVICI regimen respectively in part 1 and part 2 per cycle.
Drug: Etoposide — Participants will receive a cumulative dose of etoposide 300 mg/m^2 in part 1 and part 2 as a part of RICE regimen per cycle.
Drug: Vincristine — Participants will receive a cumulative dose of vincristine 1.6 mg/m^2 in part 1 and part 2 as a part of RVICI regimen per cycle.
Drug: Idarubicin — Participants will receive a cumulative dose of idarubicin 20 mg/m^2 in part 1 and part 2 as a part of RVICI regimen per cycle.
Drug: Dexamethasone — Participants will receive a cumulative dose of dexamethasone 100 mg/m^2 in part 1 and part 2 as a part of RICE/RVICI regimen per cycle.

SUMMARY:
The purpose of this study is to confirm that the pharmacokinetics of ibrutinib in pediatric participants is consistent with that in adults (part 1) and to assess efficacy (event-free survival [EFS]) of ibrutinib in combination with rituximab, ifosfamide, carboplatin, and etoposide (RICE) or rituximab, vincristine, ifosfamide, carboplatin, and idarubicin (RVICI) background therapy compared to RICE or RVICI background therapy alone (part 2).

DETAILED DESCRIPTION:
This is a Phase 3, randomized (study medication assigned to participants by chance), open-label (identity of study drug will be known to participant and study staff), controlled study which consists of two parts: Part 1 and Part 2. The Part 1 is a pharmacokinetic run-in part, which will be conducted before starting the randomized part (Part 2) of the study and Part 2 is a randomized and open-label study. Part 1 and Part 2 of the study will be conducted in 3 phases: a Pretreatment (Screening) Phase (Up to 14 days before administration of study drug), a Treatment Phase, and a Posttreatment Phase. The Treatment Phase will extend from enrollment (in Part 1) or randomization (in Part 2) until 1 of the following: 1) completion of 3 cycles of therapy, 2) transplantation, if clinically indicated, or 3) progressive disease (PD), whichever comes first. The Posttreatment Phase will continue until death, loss to follow up, consent withdrawal, or study end, whichever occurs first. The end of study is defined as when approximately 60 event-free survival (EFS) events have occurred in Part 2 (death, disease progression, or lack of complete response [CR] or partial response [PR] after 3 cycles of treatment based on blinded independent event review), or the sponsor terminates the study, whichever comes first. Participants in Part 1 will be 1 to less than (<) 18 years old. Participants in Part 2 will be 1 to 30 years old. Participants will be primarily evaluated for pharmacokinetics in part 1 and efficacy (EFS) of ibrutinib in combination with RICE or RVICI background therapy compared to RICE or RVICI background therapy alone in part 2. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with 1 to less than (<) 18 years of age (Part 1 only), or 1 to 30 years of age, inclusive, if initial diagnosis of mature B-cell non-Hodgkin lymphoma (NHL) occurred at <18 years of age (Part 2 only)
* Participants must be in first recurrence and have received only one prior line of therapy or have disease that is primarily refractory to conventional therapy
* Participants must have at least 1 of the following: 1 site of measurable disease greater than (>) 1 centimeter (cm) in the longest diameter and >1 cm in the shortest diameter by radiological imaging; bone marrow involvement; cerebrospinal fluid with blasts present
* Participants with lansky-Karnofsky score of greater than or equal to (>=) 50
* Adolescent women/young women of childbearing potential must have a negative highly sensitive serum or urine beta-human chorionic gonadotropin (beta-hCG) pregnancy test at Screening before enrollment/randomization. Adolescent/young women who are pregnant or breastfeeding are ineligible for this study

Exclusion Criteria:

* Participants with ongoing anticoagulation treatment with warfarin or equivalent vitamin K antagonists (example phenprocoumon), or ongoing treatment with agents known to be strong CYP3A4/5 inhibitors, or has taken any disallowed therapies as noted in Section 8.2, Prohibited Medications, before the planned first dose of study drug
* Participants with inherited or acquired bleeding disorders
* Participants with clinically significant arrhythmias, complex congenital heart disease, or left ventricular ejection fraction (LVEF) <50 percent (%) or shortening fraction (SF) <=28%
* Participants with known history of human immunodeficiency virus (HIV) or active Hepatitis B or C virus
* Participants with any condition that could interfere with the absorption or metabolism of ibrutinib including malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel
* Participants with known allergies, hypersensitivity, or intolerance to ibrutinib or its excipients (refer to Investigator's Brochure)
* A diagnosis of post-transplant lymphoproliferative disease (PTLD)
* Participants who are within 6 months of an allogeneic bone marrow transplant
* Participants who have had prior exposure to ibrutinib

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (76):
- United States (17):
  - Los Angeles, California
  - Orange, California
  - Palo Alto, California
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Atlanta, Georgia
  - Baltimore, Maryland
  - Boston, Massachusetts
  - New York, New York
  - Valhalla, New York
  - Charlotte, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Dallas, Texas
  - Salt Lake City, Utah
  - Milwaukee, Wisconsin
- Belgium (2):
  - Brussels
  - Leuven
- Brazil (3):
  - Barretos
  - Curitiba
  - São Paulo
- Bulgaria (2):
  - Plovdiv
  - Sofia
- Canada (2):
  - Halifax, Nova Scotia
  - Toronto, Ontario
- Czechia (2):
  - Brno
  - Prague
- France (8):
  - Bordeaux
  - Lille
  - Lyon
  - Marseille
  - Nantes
  - Toulouse
  - Vandœuvre-lès-Nancy
  - Villejuif
- Germany (5):
  - Berlin
  - Freiburg im Breisgau
  - Kiel
  - München
  - Münster
- Hungary (2):
  - Budapest
  - Debrecen
- Netherlands (2):
  - Rotterdam
  - Utrecht
- Poland (3):
  - Krakow
  - Warsaw
  - Wroclaw
- Romania (4):
  - Bucharest
  - Cluj-Napoca
  - Oradea
  - Timișoara
- Russia (3):
  - Moscow
  - Saint Petersburg
  - Yekaterinburg
- Seoul, South Korea
- Spain (4):
  - Barcelona
  - Esplugues de Llobregat
  - Madrid
  - Valencia
- Gothenburg, Sweden
- Taiwan (3):
  - Kaohsiung City
  - Taipei
  - Taoyuan District
- Turkey (Türkiye) (2):
  - Ankara
  - Izmir
- Kiev, Ukraine
- United Kingdom (9):
  - Birmingham
  - Cambridge
  - Leeds
  - Liverpool
  - London
  - Manchester
  - Newcastle
  - Sheffield
  - Surrey

REFERENCES:
- [Derived] Burke GAA, Vinti L, Kabickova E, Beishuizen A, Tacyildiz N, Uyttebroeck A, Kang HJ, Luisi F, Minard-Colin V, Burkhardt B, Tamegnon M, Sun S, Curtis M, Deshpande S, Nottage K, Howes A, Srinivasan S, Bhojwani D, Norris R, Cairo M. Ibrutinib plus RICE or RVICI for relapsed/refractory mature B-cell non-Hodgkin lymphoma in children and young adults: SPARKLE trial. Blood Adv. 2023 Feb 28;7(4):602-610. doi: 10.1182/bloodadvances.2022008802. PMID 36541957
- [Derived] Chu Y, Lee S, Shah T, Yin C, Barth M, Miles RR, Ayello J, Morris E, Harrison L, Van de Ven C, Galardy P, Goldman SC, Lim MS, Hermiston M, McAllister-Lucas LM, Giulino-Roth L, Perkins SL, Cairo MS. Ibrutinib significantly inhibited Bruton's tyrosine kinase (BTK) phosphorylation,in-vitro proliferation and enhanced overall survival in a preclinical Burkitt lymphoma (BL) model. Oncoimmunology. 2018 Oct 11;8(1):e1512455. doi: 10.1080/2162402X.2018.1512455. eCollection 2019. PMID 30546948

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1: Ibrutinib+RICE: Participants received ibrutinib based on age group and body surface area (BSA) in combination with chemoimmunotherapy (CIT) (investigator choice of RICE [rituximab, ifosfamide, carboplatin, etoposide, and dexamethasone]). For both regimens, triple intrathecal therapy consisting of methotrexate, corticosteroid, and cytarabine will be administered for central nervous system (CNS) prophylaxis in age-appropriate dosing. Ibrutinib suspension or capsule was administered once daily starting Day 1 Cycle 1. The first 2 participants enrolled in each age group (1-5 years, 6-11 years, and 12-17 years) received Ibrutinib at a lower starting dose of 240 milligram per meter square (mg/m^2) (not to exceed 420 mg per day) for the first cycle (older children [6-17 years] were enrolled first before enrolling younger children [1-5 years]), followed by dose escalation to 329 mg/m^2 (not to exceed 560 mg per day) at the start of Cycle 2 based on the safety assessments. The RICE regimen was composed of rituximab 750 mg/m^2, ifosfamide 9 grams per meter square (g/m^2), carboplatin 635 mg/m^2, etoposide 300 mg/m^2, and dexamethasone 100 mg/m^2. Study treatment continued for 3 cycles (each cycle of 28 or 21 days), unless the participants experienced unacceptable toxicity or disease progression.
- Part 1: Ibrutinib+RVICI: Participants received ibrutinib based on age group and BSA in combination with CIT (investigator choice of RVICI [rituximab, vincristine, ifosfamide, carboplatin, idarubicin, and dexamethasone]). dexamethasone]). For both regimens, triple intrathecal therapy consisting of methotrexate, corticosteroid, and cytarabine will be administered for central nervous system (CNS) prophylaxis in age-appropriate dosing. The first 2 participants enrolled in each age group (1-5 years, 6-11 years, and 12-17 years) received Ibrutinib at a lower starting dose of 240 mg/m2 (not to exceed 420 mg per day) for the first cycle (older children [6-17 years] were enrolled first before enrolling younger children [1-5 years]), followed by dose escalation to 329 mg/m2 (not to exceed 560 mg per day) at the start of Cycle 2 based on the safety assessments. The RVICI regimen was composed of rituximab 750 mg/m^2, vincristine 1.6 mg/m^2, ifosfamide 10 g/m^2, carboplatin 800 mg/m^2, idarubicin 20 mg/m^2, and dexamethasone 100 mg/m^2. Study treatment continued for 3 cycles (each cycle of 28 or 21 days), unless the participants experienced unacceptable toxicity or disease progression.
- Part 2: Ibrutinib+CIT (RICE or RVICI): Participants received ibrutinib based on age group and BSA in combination with CIT (investigator choice of RICE or RVICI) until 3 treatment cycles, transplantation if indicated, or until progressive disease (PD) or unacceptable toxicity. For both regimens, triple intrathecal therapy consisting of methotrexate, corticosteroid, and cytarabine will be administered for central nervous system (CNS) prophylaxis in age-appropriate dosing. Participants of age groups 1-5 years and 6-11 years received ibrutinib 440 mg/m^2, and age group 12-17 years received Ibrutinib 329 mg/m^2 (dose selected from Part 1).
- Part 2: Chemoimmunotherapy: Participants received CIT (investigator choice of RICE or RVICI) alone based on age group and BSA until 3 treatment cycles, transplantation if indicated, or until PD or unacceptable toxicity. For both regimens, triple intrathecal therapy consisting of methotrexate, corticosteroid, and cytarabine will be administered for CNS prophylaxis in age-appropriate dosing. The RICE regimen was composed of rituximab 750 mg/m^2, ifosfamide 9 g/m2, carboplatin 635 mg/m^2, etoposide 300 mg/m^2, and dexamethasone 100 mg/m^2. The RVICI regimen was composed of rituximab 750 mg/m^2, vincristine 1.6 mg/m^2, idarubicin 20 mg/m^2, carboplatin 800 mg/m^2, ifosfamide 10 g/m^2, and dexamethasone 100 mg/m^2 (all doses represented as cumulative administered in 1 cycle).
Period: Overall Study
Arm/Group | Part 1: Ibrutinib+RICE | Part 1: Ibrutinib+RVICI | Part 2: Ibrutinib+CIT (RICE or RVICI) | Part 2: Chemoimmunotherapy
Started | 11 | 10 | 35 | 16
Completed | 0 | 0 | 0 | 0
Not Completed | 11 | 10 | 35 | 16
Not completed — Death | 4 | 9 | 19 | 10
Not completed — Withdrawal by Subject | 0 | 0 | 4 | 2
Not completed — Study Terminated by Sponsor | 6 | 1 | 12 | 4
Not completed — Other | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Ibrutinib+RICE | Part 1: Ibrutinib+RVICI | Part 2: Ibrutinib+CIT (RICE or RVICI) | Part 2: Chemoimmunotherapy | Total
Number analyzed (Participants) | 11 | 10 | 35 | 16 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.5 (4.91) | 8.3 (3.43) | 13.9 (3.94) | 13.2 (4.37) | 12.4 (4.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 12 | 3 | 19
  Male | 8 | 9 | 23 | 13 | 53
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 8 | 6 | 15
  Black or African American | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  White | 9 | 10 | 22 | 8 | 49
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 3 | 0 | 4
  Other | 0 | 0 | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  BELGIUM | 0 | 0 | 2 | 0 | 2
  BRAZIL | 1 | 0 | 1 | 2 | 4
  BULGARIA | 0 | 0 | 2 | 0 | 2
  CANADA | 0 | 0 | 1 | 0 | 1
  CZECH REPUBLIC | 0 | 2 | 2 | 0 | 4
  FRANCE | 2 | 1 | 3 | 1 | 7
  GERMANY | 2 | 1 | 3 | 0 | 6
  ITALY | 2 | 1 | 4 | 2 | 9
  NETHERLANDS | 0 | 0 | 1 | 1 | 2
  POLAND | 0 | 1 | 0 | 2 | 3
  ROMANIA | 1 | 0 | 0 | 0 | 1
  RUSSIAN FEDERATION | 0 | 0 | 2 | 0 | 2
  SOUTH KOREA | 1 | 0 | 5 | 4 | 10
  SPAIN | 0 | 0 | 2 | 0 | 2
  SWEDEN | 0 | 0 | 1 | 0 | 1
  TAIWAN | 0 | 0 | 2 | 1 | 3
  TURKEY | 1 | 4 | 1 | 2 | 8
  UKRAINE | 0 | 0 | 1 | 0 | 1
  UNITED KINGDOM | 0 | 0 | 1 | 1 | 2
  UNITED STATES | 1 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Area Under the Plasma Concentration-time Curve (AUC) of Ibrutinib
Description: AUC is defined as area under the plasma concentration-time curve. As per planned analyses, pharmacokinetic (PK) parameters for Part 1 were presented per dose group (240 milligrams per meter square [mg/m^2], 329 mg/m^2 and 440 mg/m^2) and age group (1-5, 6-11, 12-17 and >18 years). As planned in protocol, the PK parameters were presented per dose group as dosing was dependent on age.
Time Frame: Up to Cycle 3 (each cycle of 21 or 28 days)
Population: PK analysis set included participants in the ibrutinib group that received ibrutinib doses and had quantifiable plasma concentration of ibrutinib. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure. Here, "n (number analyzed)" is defined as number of participants analyzed for specified category.
Measure: Median (Full Range); unit: hours*nanogram per milliliter (h*ng/mL)
Groups:
- Part 1: Ibrutinib: 240 mg/m^2: Participants received 240 milligrams per meter square (mg/m^2) ibrutinib based on age group for 3 treatment cycles with each cycle of 21 or 28 days long in Part 1.
- Part 1: Ibrutinib: 329 mg/m^2: Participants received 329 mg/m^2 ibrutinib based on age group for 3 treatment cycles with each cycle of 21 or 28 days long in Part 1.
- Part 1: Ibrutinib: 440 mg/m^2: Participants received 440 mg/m^2 ibrutinib based on age group for 3 treatment cycles with each cycle of 21 or 28 days long in Part 1.
Arm/Group | Part 1: Ibrutinib: 240 mg/m^2 | Part 1: Ibrutinib: 329 mg/m^2 | Part 1: Ibrutinib: 440 mg/m^2
Number analyzed (Participants) | 3 | 10 | 7
hours*nanogram per milliliter (h*ng/mL)
  1-5 years: number analyzed (Participants) | 2 | 1 | 3
  1-5 years | 143 [116 to 170] | 386 [386 to 386] | 310 [230 to 543]
  6-11 years | 145 [140 to 233] | 349 [238 to 562] | 324 [185 to 538]
  12-17 years: number analyzed (Participants) | 3 | 8 | 0
  12-17 years | 1210 [939 to 1450] | 661 [394 to 778] |
  18+ years: number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Part 1: Apparent (Oral) Plasma Clearance (CL/F) of Ibrutinib
Description: CL/F is defined as apparent plasma clearance of ibrutinib. As per planned analyses, PK parameters for Part 1 were presented per dose group (240 mg/m^2, 329 mg/m^2 and 440 mg/m^2) and age group (1-5, 6-11, 12-17 and >18 years). As planned in protocol, the PK parameters were presented per dose group as dosing was dependent on age.
Time Frame: Up to Cycle 3 (each cycle of 21 or 28 days)
Population: as for outcome 1
Measure: Median (Full Range); unit: milliliter per hour (mL/h)
Arm/Group | Part 1: Ibrutinib: 240 mg/m^2 | Part 1: Ibrutinib: 329 mg/m^2 | Part 1: Ibrutinib: 440 mg/m^2
Number analyzed (Participants) | 3 | 10 | 7
milliliter per hour (mL/h)
  1-5 years: number analyzed (Participants) | 2 | 1 | 3
  1-5 years | 1220 [1000 to 1430] | 508 [508 to 508] | 1200 [838 to 1550]
  6-11 years | 1450 [1080 to 1500] | 805 [664 to 1100] | 1300 [910 to 2460]
  12-17 years: number analyzed (Participants) | 3 | 8 | 0
  12-17 years | 348 [340 to 433] | 729 [568 to 1330] |
  18+ years: number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Part 1: Apparent (Oral) Volume of Distribution (Vd/F) of Ibrutinib
Description: Vd/F is defined as apparent (oral) volume of distribution of ibrutinib. As per planned analyses, pharmacokinetic (PK) parameters for Part 1 were presented per dose group (240 mg/m^2, 329 mg/m^2 and 440 mg/m^2) and age group (1-5, 6-11, 12-17 and >18 years). As planned in protocol, the PK parameters were presented per dose group as dosing was dependent on age.
Time Frame: Up to Cycle 3 (each cycle of 21 or 28 days)
Population: PK analysis set included participants in the ibrutinib group that received ibrutinib doses and had quantifiable plasma concentration of ibrutinib. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure. Here, n (number analyzed)" is defined as number of participants analyzed for specified category.
Measure: Median (Full Range); unit: liter(s)
Arm/Group | Part 1: Ibrutinib: 240 mg/m^2 | Part 1: Ibrutinib: 329 mg/m^2 | Part 1: Ibrutinib: 440 mg/m^2
Number analyzed (Participants) | 3 | 10 | 7
liter(s)
  1-5 years: number analyzed (Participants) | 2 | 1 | 3
  1-5 years | 11.1 [8.26 to 13.9] | 5.18 [5.18 to 5.18] | 7.63 [5.34 to 11.1]
  6-11 years | 18 [10.8 to 29.9] | 7.55 [2.89 to 15.6] | 19 [6.09 to 55.9]
  12-17 years: number analyzed (Participants) | 3 | 8 | 0
  12-17 years | 3.63 [2.32 to 4.77] | 11.3 [6.34 to 18.5] |
  18+ years: number analyzed (Participants) | 0 | 0 | 0

4. Primary Outcome: Part 1: Maximum Observed Plasma Concentration (Cmax) of Ibrutinib
Description: Cmax is defined as maximum plasma concentration of ibrutinib. As per planned analyses, pharmacokinetic (PK) parameters for Part 1 were presented per dose group (240 mg/m^2, 329 mg/m^2 and 440 mg/m^2) and age group (1-5, 6-11, 12-17 and >18 years). As planned in protocol, the PK parameters were presented per dose group as dosing was dependent on age.
Time Frame: Up to Cycle 3 (each cycle of 21 or 28 days)
Population: as for outcome 1
Measure: Median (Full Range); unit: nanograms per milliliter (ng/mL)
Arm/Group | Part 1: Ibrutinib: 240 mg/m^2 | Part 1: Ibrutinib: 329 mg/m^2 | Part 1: Ibrutinib: 440 mg/m^2
Number analyzed (Participants) | 3 | 10 | 7
nanograms per milliliter (ng/mL)
  1-5 years: number analyzed (Participants) | 2 | 1 | 3
  1-5 years | 3.86 [3.75 to 3.98] | 4.48 [4.48 to 4.48] | 5.07 [4.5 to 5.14]
  6-11 years | 3.46 [3.12 to 3.6] | 3.64 [3.32 to 4.59] | 3.88 [3.2 to 4.44]
  12-17 years: number analyzed (Participants) | 3 | 8 | 0
  12-17 years | 4.88 [4.76 to 5.4] | 4.73 [4.07 to 5.07] |
  18+ years: number analyzed (Participants) | 0 | 0 | 0

5. Primary Outcome: Part 1: Relationship Between AUC and Body Size
Description: The relationship between ibrutinib metrics of systemic exposure (AUC) with body size was assessed to determine the impact on AUC which were presented per dose groups (240 mg/m^2, 329 mg/m^2 and 440 mg/m^2) and age groups (1-5, 6-11, 12-17 and >18 years). The data could not be analyzed in tabular format for this outcome measure as they correspond to a flat regression line in nonlinear mixed effects modeling.
Time Frame: Up to Cycle 3 (each cycle of 28 days)
Population: PK analysis set included participants in the ibrutinib group that received ibrutinib doses and had quantifiable plasma concentration of ibrutinib.
Arm/Group | Part 1: Ibrutinib+RICE | Part 1: Ibrutinib+RVICI
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Part 2: Event Free Survival (EFS) Between the 2 Treatment Groups
Description: EFS was the time interval from randomization to death, disease progression, or lack of complete response (CR) or partial response (PR) after 3 cycles of treatment, whichever occurred first based on blinded independent event review by the Independent Review Committee (IRC). CR was defined as computed tomography (CT) or magnetic resonance imaging (MRI) reveals no residual disease or new lesions, resected residual mass that was pathologically (morphologically) negative for disease, BM and CSF morphologically free of disease with no new lesions by imaging examination. PR was defined as 50 percent (%) decrease in sum of the products of the lesion diameters (SPD) on CT or MRI; fluorodeoxyglucose (FDG)-positron emission tomography (PET) may be positive, no new or progressive disease (PD); morphologic evidence of disease may be present in BM or cerebrospinal fluid (CSF) if present at diagnosis; however, there should be 50% reduction in percentage of lymphoma cells.
Time Frame: Time from Randomization to death, disease progression, or lack of CR or PR after 3 cycles of treatment (up to 4 year and 4 months)
Population: The intent-to-treat (ITT) population consisted of all randomized participants; participants analyzed based on randomization, regardless of study drug received. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2: Ibrutinib+CIT (RICE or RVICI) | Part 2: Chemoimmunotherapy
Number analyzed (Participants) | 35 | 16
Months | 6.05 [2.99 to 8.84] | 6.97 [2.60 to 11.07]

7. Secondary Outcome: Part 1 and Part 2: Number of Participants With Adverse Events as Measure of Safety and Tolerability
Description: An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Time Frame: Up to 4 year and 4 months
Population: Safety population consisted of all participants who received at least 1 dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Ibrutinib+RICE | Part 1: Ibrutinib+RVICI | Part 2: Ibrutinib+CIT (RICE or RVICI) | Part 2: Chemoimmunotherapy
Number analyzed (Participants) | 11 | 10 | 35 | 15
Participants | 11 | 10 | 35 | 15

8. Secondary Outcome: Part 1 and Part 2: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants achieving a best overall response of either complete response (CR) (including CR biopsy-negative [CRb] and unconfirmed CR [CRu]) or partial response (PR) as evaluated by International Pediatric non-Hodgkin lymphoma (NHL) response criteria. CR=disappearance of all disease; CRb=residual mass has no morphologic evidence of disease from limited or core biopsy, with no new lesions by imaging examination; bone marrow (BM) and CSF morphologically free of disease; no new or PD elsewhere, CRu=Residual mass is negative by FDG-PET; no new lesions by imaging examination; BM and CSF morphologically free of disease; no new or PD elsewhere, PR=50% decrease in SPD on CT or MRI; FDG-PET may be positive (deauville score or 4 or 5 with reduced lesional uptake compared with baseline); no new or PD; morphologic evidence of disease may be present in BM or CSF if present at diagnosis; however, there should be 50% reduction in percentage of lymphoma cells.
Time Frame: Up to 4 year and 4 months
Population: The ITT Population consisted of all randomized participants; participants analyzed based on randomization, regardless of study drug received.
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: Ibrutinib+RICE | Part 1: Ibrutinib+RVICI | Part 2: Ibrutinib+CIT (RICE or RVICI) | Part 2: Chemoimmunotherapy
Number analyzed (Participants) | 11 | 10 | 35 | 16
Percentage of participants | 81.8 | 50.0 | 68.6 | 81.3

9. Secondary Outcome: Part 1 and Part 2: Gene Expression Evaluated by Disease-specific Biomarkers at Baseline
Description: Tumor formalin-fixed paraffin-embedded (FFPE) samples were taken to evaluate the baseline gene expression by disease-specific biomarkers such as BCL-2L1 (BCL-xl), BIRC2 (cIAP1), Caspase 3 (CASP3), STAT3, and SYK. Transcripts per million (TPM) is a normalization method for RNA-sequencing, which means "for every 1,000,000 RNA molecules in the RNA-sequencing tumor FFPE sample, x came from this gene/transcript.
Time Frame: Baseline
Population: Biomarker analyses were conducted on the ITT population. As per change in planned analysis, genetic analysis was not performed for Part 1. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Transcripts per million
Arm/Group | Part 1: Ibrutinib+RICE | Part 1: Ibrutinib+RVICI | Part 2: Ibrutinib+CIT (RICE or RVICI) | Part 2: Chemoimmunotherapy
Number analyzed (Participants) | 0 | 0 | 18 | 9
Transcripts per million
  BCL-2L1 (BCL-xl) |  |  | 58.09346 (38.75996) | 74.30790 (75.82331)
  BIRC2 (cIAP1) |  |  | 47.20787 (16.26430) | 40.01716 (9.28104)
  Caspase 3 (CASP3) |  |  | 51.14711 (21.44109) | 47.61412 (32.12666)
  STAT3 |  |  | 540.02256 (363.75256) | 526.35308 (473.08255)
  SYK |  |  | 705.29909 (503.07085) | 618.36324 (144.72067)

10. Secondary Outcome: Part 1 and Part 2: Number of Participants With Immunoglobulin and T-cell Receptor Gene Rearrangements
Description: Number of participants with immunoglobulin and T-cell receptor gene rearrangements were reported.
Time Frame: At baseline (Cycle 1 Day 1) of Part 1 and 2
Population: Biomarker analyses were conducted on the ITT population. As per change in planned analysis, immunoglobulin and T-cell receptor gene rearrangements were not performed for Part 1 and Part 2.
Arm/Group | Part 1: Ibrutinib+RICE | Part 1: Ibrutinib+RVICI | Part 2: Ibrutinib+CIT (RICE or RVICI) | Part 2: Chemoimmunotherapy
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Part 1 and Part 2: Number of Participants With Greater Than (>) 90% Bruton's Tyrosine Kinase (BTK) Occupancy
Description: Number of participants with >90% BTK occupancy were reported. Blood samples were collected to assess BTK occupancy.
Time Frame: Up to 3 months
Population: Biomarker analyses were conducted on the ITT population. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure. As planned, BTK occupancy was assessed for ibrutinib only.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Ibrutinib: Participants received ibrutinib based on age group and body surface area (BSA) in combination with chemoimmunotherapy (CIT) (investigator choice of RICE [rituximab, ifosfamide, carboplatin, etoposide, and dexamethasone]). For both regimens, triple intrathecal therapy consisting of methotrexate, corticosteroid, and cytarabine will be administered for central nervous system (CNS) prophylaxis in age-appropriate dosing. Ibrutinib suspension or capsule was administered once daily starting Day 1 Cycle 1. The first 2 participants enrolled in each age group (1-5 years, 6-11 years, and 12-17 years) received Ibrutinib at a lower starting dose of 240 milligram per meter square (mg/m^2) (not to exceed 420 mg per day) for the first cycle (older children [6-17 years] were enrolled first before enrolling younger children [1-5 years]), followed by dose escalation to 329 mg/m^2 (not to exceed 560 mg per day) at the start of Cycle 2 based on the safety assessments. The RICE regimen was composed of rituximab 750 mg/m^2, ifosfamide 9 grams per meter square (g/m^2), carboplatin 635 mg/m^2, etoposide 300 mg/m^2, and dexamethasone 100 mg/m^2. Study treatment continued for 3 cycles (each cycle of 28 or 21 days), unless the participants experienced unacceptable toxicity or disease progression.
- Part 2: Ibrutinib: Participants received ibrutinib based on age group and BSA in combination with CIT (investigator choice of RVICI [rituximab, vincristine, ifosfamide, carboplatin, idarubicin, and dexamethasone]). dexamethasone]). For both regimens, triple intrathecal therapy consisting of methotrexate, corticosteroid, and cytarabine will be administered for central nervous system (CNS) prophylaxis in age-appropriate dosing. The first 2 participants enrolled in each age group (1-5 years, 6-11 years, and 12-17 years) received Ibrutinib at a lower starting dose of 240 mg/m2 (not to exceed 420 mg per day) for the first cycle (older children [6-17 years] were enrolled first before enrolling younger children [1-5 years]), followed by dose escalation to 329 mg/m2 (not to exceed 560 mg per day) at the start of Cycle 2 based on the safety assessments. The RVICI regimen was composed of rituximab 750 mg/m^2, vincristine 1.6 mg/m^2, ifosfamide 10 g/m^2, carboplatin 800 mg/m^2, idarubicin 20 mg/m^2, and dexamethasone 100 mg/m^2. Study treatment continued for 3 cycles (each cycle of 28 or 21 days), unless the participants experienced unacceptable toxicity or disease progression.
Arm/Group | Part 1: Ibrutinib | Part 2: Ibrutinib
Number analyzed (Participants) | 15 | 13
Participants | 5 | 5

12. Secondary Outcome: Part 1 and Part 2: Visual Analog Scale (VAS) Score for Palatability
Description: Palatability of ibrutinib was measured by using a VAS. The scale is a 5-point visual analog scale incorporating a facial hedonic scale designed to span pediatric ages and levels of participant comprehension with a score range of 1 to 5, where 1 represents best score and 5 is worst palatability.
Time Frame: Day 1 of Cycle 1 and Cycle 3
Population: Safety population: all participants who received at least 1 dose of treatment. Here 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure (OM) and, n (number analyzed) signifies number of participants analyzed for specified category. Participants in arm 'Part 2: Chemoimmunotherapy' did not receive ibrutinib, and palatability of ibrutinib was measured in this OM. Hence, no data available to report for this arm.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Part 1: Ibrutinib+RICE | Part 1: Ibrutinib+RVICI | Part 2: Ibrutinib+CIT (RICE or RVICI)
Number analyzed (Participants) | 11 | 10 | 32
Units on a scale
  Cycle 1 Day 1 | 2.6 (1.21) | 3.2 (1.40) | 2.4 (1.16)
  Cycle 3 Day 1: number analyzed (Participants) | 8 | 3 | 16
  Cycle 3 Day 1 | 3.3 (1.39) | 2.3 (1.15) | 2.6 (0.89)

13. Secondary Outcome: Part 1: Number of Participants With CD79B, CARD11, and MYD Mutations
Description: Number of Participants with CD79B, CARD11, and MYD Mutations were reported.
Time Frame: Up to 4 years and 4 months
Population: Biomarker analyses were conducted on the ITT population. As per change in planned analysis, genetic analysis was not performed for Part 1.
Arm/Group | Part 1: Ibrutinib+RICE | Part 1: Ibrutinib+RVICI
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Part 2: Number of Participants With CD79B, CARD11, and MYD Mutations
Description: Number of participants with CD79B, CARD11, and MYD mutations were reported. Blood samples were taken to evaluate the levels of biomarkers such as CD79B, CARD11, and MYD mutations.
Time Frame: Up to 4 year and 4 months
Population: Biomarker analyses were conducted on the ITT population. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Ibrutinib+CIT (RICE or RVICI) | Part 2: Chemoimmunotherapy
Number analyzed (Participants) | 20 | 10
Participants
  CD79B | 1 | 0
  CARD11 | 1 | 0
  MYD mutation | 0 | 0

15. Secondary Outcome: Part 1: Number of Participants With c-MYC Gene Rearrangement
Description: Number of participants with c-MYC gene rearrangement were reported.
Time Frame: At baseline (Cycle 1 Day 1)
Population: as for outcome 13
Arm/Group | Part 1: Ibrutinib+RICE | Part 1: Ibrutinib+RVICI
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Part 2: Number of Participants With c-MYC Gene Rearrangement
Description: Number of participants with c-MYC gene rearrangement were reported. Blood samples were taken to evaluate the levels of biomarker such as c-MYC Gene rearrangement.
Time Frame: At baseline (Cycle 1 Day 1)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Ibrutinib+CIT (RICE or RVICI) | Part 2: Chemoimmunotherapy
Number analyzed (Participants) | 18 | 9
Participants | 1 | 1

17. Secondary Outcome: Part 2: Percentage of Participants Who Achieved Complete Response (CR)
Description: Complete response rate was defined as the percentage of participants who achieved complete response or complete response with an incomplete marrow recovery (CRi) on or prior to initiation of subsequent anti-leukemic therapy per the IRC assessment.
Time Frame: Up to 4 year and 4 months
Population: as for outcome 8
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 2: Ibrutinib+CIT (RICE or RVICI) | Part 2: Chemoimmunotherapy
Number analyzed (Participants) | 35 | 16
Percentage of Participants | 17.1 | 18.8

18. Secondary Outcome: Part 2: Percentage of Participants Who Achieved Partial Response (PR)
Description: Percentage of participants who achieved PR were assessed. PR was defined as 50% decrease in SPD on computed tomography (CT) or magnetic resonance imaging (MRI); FDG-PET may be positive; no new or PD; morphologic evidence of disease may be present in BM or cerebrospinal fluid (CSF) if present at diagnosis; however, there should be 50% reduction in percentage of lymphoma cells.
Time Frame: Up to 4 year and 4 months
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Groups:
- Part 2: Chemoimmunotherapy: Participants received CIT (investigator choice of RICE or RVICI) alone based on age group and BSA until 3 treatment cycles, transplantation if indicated, or until PD or unacceptable toxicity. For both regimens, triple intrathecal therapy consisting of methotrexate, corticosteroid, and cytarabine will be administered for CNS prophylaxis in age-appropriate dosing. The RICE regimen was composed of rituximab 750 mg/m^2, ifosfamide 9 g/m^2, carboplatin 635 mg/m^2, etoposide 300 mg/m^2, and dexamethasone 100 mg/m^2. The RVICI regimen was composed of rituximab 750 mg/m^2, vincristine 1.6 mg/m^2, idarubicin 20 mg/m^2, carboplatin 800 mg/m^2, ifosfamide 10 g/m^2, and dexamethasone 100 mg/m^2 (all doses represented as cumulative administered in 1 cycle).
Arm/Group | Part 2: Ibrutinib+CIT (RICE or RVICI) | Part 2: Chemoimmunotherapy
Number analyzed (Participants) | 35 | 16
percentage of participants | 51.4 | 62.5

19. Secondary Outcome: Part 2: Tumor Volume Reduction Rate at Day 14
Description: The tumor volume reduction rate was defined as percent decrease in the sum of the products of the lesion diameters at Day 14. It was measured as the mean change in the sum of the products of the lesion diameters (SPD) at Day 14.
Time Frame: At Day 14
Population: The ITT Population consisted of all randomized participants; participants was analyzed based on randomization, regardless of study drug received. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Deviation); unit: Percent change
Arm/Group | Part 2: Ibrutinib+CIT (RICE or RVICI) | Part 2: Chemoimmunotherapy
Number analyzed (Participants) | 30 | 11
Percent change | -49.7 (33.41) | -58.60 (34.04)

20. Secondary Outcome: Part 2: Number of Participants Who Proceeded to Stem Cell Transplantation
Description: Number of participants who proceeded to stem cell transplantation were reported.
Time Frame: Up to end of the study (Up to 4 year and 4 months)
Population: The ITT population consisted of all randomized participants; participants were analyzed based on randomization, regardless of study drug received.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Ibrutinib+CIT (RICE or RVICI) | Part 2: Chemoimmunotherapy
Number analyzed (Participants) | 35 | 16
Participants | 13 | 7

21. Secondary Outcome: Part 2: Time to Response
Description: Time to response was defined as the time interval from the first dose of ibrutinib to the first documented response for those participants who responded. Time to response was summarized for participants who achieved either CR (including CRb and CRu) or PR. CR=disappearance of all disease; CRb=residual mass has no morphologic evidence of disease from limited or core biopsy, with no new lesions by imaging examination; BM and CSF morphologically free of disease; no new or PD elsewhere, CRu=Residual mass is negative by FDG-PET; no new lesions by imaging examination; BM and CSF morphologically free of disease; no new or PD elsewhere, PR=50% decrease in SPD on CT or MRI; FDG-PET may be positive (deauville score or 4 or 5 with reduced lesional uptake compared with baseline); no new or PD; morphologic evidence of disease may be present in BM or CSF if present at diagnosis; however, there should be 50% reduction in percentage of lymphoma cells.
Time Frame: Up to 4 Years and 4 months
Population: Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure. Time to response was summarized for participants who achieved either CR (including CRb and CRu) or PR.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Part 2: Ibrutinib+CIT (RICE or RVICI) | Part 2: Chemoimmunotherapy
Number analyzed (Participants) | 24 | 13
Months | 0.89 [0.49 to 1.87] | 0.82 [0.46 to 1.94]

22. Secondary Outcome: Part 2: Duration of Response
Description: Duration of response was defined as the duration from date of initial documentation of a response (CR or PR) to the date of first documented evidence of progressive disease (PD) or death, whichever occurred first. PD: >25% increase in SPD of residual lesions (calculated from nadir) on CT or MRI; Deauville score 4 or 5 on FDG-PET with increase in lesional uptake from baseline; documentation of new lesions or development of new morphologic evidence of disease in BM or CSF.
Time Frame: Up to 4 year and 4 months
Population: Duration of response was summarized for participants who achieved either CR (including CRb and CRu) or PR. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Part 2: Ibrutinib+CIT (RICE or RVICI) | Part 2: Chemoimmunotherapy
Number analyzed (Participants) | 24 | 13
Months | 6.01 [3.06 to NA] — Here "NA" indicates that upper limit of 90% confidence interval was not estimable due to insufficient number of events. | 6.51 [4.53 to 10.64]

23. Secondary Outcome: Part 2: Percentage of Participants With EFS at 2 Years
Description: EFS was the time interval from randomization to death, disease progression, or lack of complete response (CR) or partial response (PR) after 3 cycles of treatment, whichever occurred first based on blinded independent event review by the IRC. CR was defined as CT or MRI reveals no residual disease or new lesions, resected residual mass that is pathologically (morphologically) negative for disease, BM and CSF morphologically free of disease with no new lesions by imaging examination. PR was defined as 50% decrease in um of the products of the SPD on CT or MRI; FDG-PET may be positive, no new or PD; morphologic evidence of disease may be present in BM or CSF if present at diagnosis; however, there should be 50% reduction in percentage of lymphoma cells.
Time Frame: At 2 years
Population: as for outcome 20
Measure: Number; unit: Percentage of participants
Arm/Group | Part 2: Ibrutinib+CIT (RICE or RVICI) | Part 2: Chemoimmunotherapy
Number analyzed (Participants) | 35 | 16
Percentage of participants | 14.3 | 12.5

24. Secondary Outcome: Part 2: Percentage of Participants With EFS at 3 Years
Description: EFS is the time interval from randomization to death, disease progression, or lack of complete response (CR) or partial response (PR) after 3 cycles of treatment, whichever occurs first based on blinded independent event review by the IRC. CR was defined as CT or MRI reveals no residual disease or new lesions, resected residual mass that is pathologically (morphologically) negative for disease, BM and CSF morphologically free of disease with no new lesions by imaging examination. PR was defined as 50% decrease in um of the products of the SPD on CT or MRI; FDG-PET may be positive, no new or PD; morphologic evidence of disease may be present in BM or CSF if present at diagnosis; however, there should be 50% reduction in percentage of lymphoma cells.
Time Frame: At 3 years
Population: as for outcome 20
Measure: Number; unit: Percentage of participants
Arm/Group | Part 2: Ibrutinib+CIT (RICE or RVICI) | Part 2: Chemoimmunotherapy
Number analyzed (Participants) | 35 | 16
Percentage of participants | 8.6 | 12.5

25. Secondary Outcome: Part 2: Overall Survival
Description: Overall survival was defined as duration from the date of randomization to the date of the participant's death.
Time Frame: Up to 4 year and 4 months
Population: as for outcome 20
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Part 2: Ibrutinib+CIT (RICE or RVICI) | Part 2: Chemoimmunotherapy
Number analyzed (Participants) | 35 | 16
Months | 14.13 [5.98 to NA] — Here "NA" indicates that upper limit of 90% Confidence interval was not estimable due to insufficient number of participants with events. | 11.07 [7.39 to NA] — Here "NA" indicates that upper limit of 90% Confidence interval was not estimable due to insufficient number of participants with events.

26. Secondary Outcome: Part 2: Area Under the Plasma Concentration-time Curve (AUC) of Ibrutinib
Description: AUC is defined as area under the plasma concentration-time curve. As per planned analyses, PK parameters for Part 2 were presented per dose group (240 mg/m^2, 329 mg/m^2 and 440 mg/m^2) and age group (1-5, 6-11, 12-17 and >18 years). As planned in protocol, the PK parameters were presented per dose group as dosing was dependent on age.
Time Frame: Up to Cycle 3 (each cycle of 21 or 28 days)
Population: as for outcome 1
Measure: Mean (Full Range); unit: h*ng/mL
Groups:
- Part 2: Ibrutinib: 240 mg/m^2:: Participants received 240 milligrams per meter square (mg/m^2) ibrutinib based on age group for 3 treatment cycles with each cycle of 21 or 28 days long in part 2.
- Part 2: Ibrutinib: 329 mg/m^2: Participants received 329 mg/m^2 ibrutinib based on age group for 3 treatment cycles with each cycle of 21 or 28 days long in part 2.
- Part 2: Ibrutinib: 440 mg/m^2: Participants received 440 mg/m^2 ibrutinib based on age group for 3 treatment cycles with each cycle of 21 or 28 days long in part 2.
Arm/Group | Part 2: Ibrutinib: 240 mg/m^2: | Part 2: Ibrutinib: 329 mg/m^2 | Part 2: Ibrutinib: 440 mg/m^2
Number analyzed (Participants) | 1 | 19 | 3
h*ng/mL
  1-5 years: number analyzed (Participants) | 0 | 0 | 2
  1-5 years |  |  | 298 [268 to 327]
  6-11 years: number analyzed (Participants) | 0 | 0 | 3
  6-11 years |  |  | 655 [428 to 879]
  12-17 years: number analyzed (Participants) | 1 | 19 | 0
  12-17 years | 215 [215 to 215] | 499 [262 to 887] |
  18+ years: number analyzed (Participants) | 0 | 2 | 0
  18+ years |  | 423 [348 to 498] |

27. Secondary Outcome: Part 2: Apparent (Oral) Plasma Clearance (CL/F) of Ibrutinib
Description: CL/F is defined as apparent plasma clearance of ibrutinib. As per planned analyses, PK parameters for Part 2 were presented per dose group (240 mg/m^2, 329 mg/m^2 and 440 mg/m^2) and age group (1-5, 6-11, 12-17 and >18 years). As planned in protocol, the PK parameters were presented per dose group as dosing was dependent on age.
Time Frame: Up to Cycle 3 (each cycle of 21 or 28 days)
Population: as for outcome 1
Measure: Median (Full Range); unit: mL/h
Groups:
- Part 2: Ibrutinib: 240 mg/m^2: Participants received 240 milligrams per meter square (mg/m^2) ibrutinib based on age group for 3 treatment cycles with each cycle of 21 or 28 days long in Part 2.
Arm/Group | Part 2: Ibrutinib: 240 mg/m^2 | Part 2: Ibrutinib: 329 mg/m^2 | Part 2: Ibrutinib: 440 mg/m^2
Number analyzed (Participants) | 1 | 19 | 3
mL/h
  1-5 years: number analyzed (Participants) | 0 | 0 | 2
  1-5 years |  |  | 1110 [1020 to 1200]
  6-11 years: number analyzed (Participants) | 0 | 0 | 3
  6-11 years |  |  | 856 [618 to 1140]
  12-17 years: number analyzed (Participants) | 1 | 19 | 0
  12-17 years | 1730 [1730 to 1730] | 982 [598 to 2010] |
  18+ years: number analyzed (Participants) | 0 | 2 | 0
  18+ years |  | 1510 [1250 to 1780] |

28. Secondary Outcome: Part 2: Apparent (Oral) Volume of Distribution (Vd/F) of Ibrutinib
Description: Vd/F is defined as apparent (oral) volume of distribution of ibrutinib. As per planned analyses, PK parameters for Part 2 were presented per dose group (240 mg/m^2, 329 mg/m^2 and 440 mg/m^2) and age group (1-5, 6-11, 12-17 and >18 years). As planned in protocol, the PK parameters were presented per dose group as dosing was dependent on age.
Time Frame: Up to Cycle 3 (each cycle of 21 or 28 days)
Population: as for outcome 1
Measure: Median (Full Range); unit: liter(s)
Arm/Group | Part 2: Ibrutinib: 240 mg/m^2 | Part 2: Ibrutinib: 329 mg/m^2 | Part 2: Ibrutinib: 440 mg/m^2
Number analyzed (Participants) | 1 | 19 | 3
liter(s)
  1-5 years: number analyzed (Participants) | 0 | 0 | 2
  1-5 years |  |  | 1.68 [1.46 to 1.91]
  6-11 years: number analyzed (Participants) | 0 | 0 | 3
  6-11 years |  |  | 6.18 [3.67 to 10.01]
  12-17 years: number analyzed (Participants) | 1 | 19 | 0
  12-17 years | 9.9 [9.9 to 9.9] | 4.14 [1.46 to 8.51] |
  18+ years: number analyzed (Participants) | 0 | 2 | 0
  18+ years |  | 9.29 [7.75 to 10.8] |

29. Secondary Outcome: Part 2: Maximum Observed Plasma Concentration (Cmax) of Ibrutinib
Description: Cmax is defined as maximum plasma concentration of ibrutinib. As per planned analyses, PK parameters for Part 2 were presented per dose group (240 mg/m^2, 329 mg/m^2 and 440 mg/m^2) and age group (1-5, 6-11, 12-17 and >18 years). As planned in protocol, the PK parameters were presented per dose group as dosing was dependent on age.
Time Frame: Up to Cycle 3 (each cycle of 21 or 28 days)
Population: as for outcome 1
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Part 2: Ibrutinib: 240 mg/m^2 | Part 2: Ibrutinib: 329 mg/m^2 | Part 2: Ibrutinib: 440 mg/m^2
Number analyzed (Participants) | 1 | 19 | 3
ng/mL
  1-5 years: number analyzed (Participants) | 0 | 0 | 2
  1-5 years |  |  | 3.79 [3.52 to 4.06]
  6-11 years: number analyzed (Participants) | 0 | 0 | 3
  6-11 years |  |  | 4.15 [3.44 to 5.01]
  12-17 years: number analyzed (Participants) | 1 | 19 | 0
  12-17 years | 2.93 [2.93 to 2.93] | 4.86 [3.12 to 5.26] |
  18+ years: number analyzed (Participants) | 0 | 2 | 0
  18+ years |  | 3.7 [3.46 to 3.94] |

30. Secondary Outcome: Part 2: Relationship Between AUC and Body Size
Description: The relationship between ibrutinib metrics of systemic exposure (AUC) with body size was assessed to determine the impact on AUC which were presented per dose groups (240 mg/m^2, 329 mg/m^2 and 440 mg/m^2) and age groups (1-5, 6-11, 12-17 and >18 years). The data could not be analyzed in tabular format for this outcome measure as they correspond to a flat regression line in nonlinear mixed effects modeling. This outcome measure was planned to be analyzed for specified arm only.
Time Frame: Up to Cycle 3 (each cycle of 28 days)
Population: as for outcome 5
Arm/Group | Part 2: Ibrutinib+CIT (RICE or RVICI)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 4 year and 4 months
Description: The safety population consisted of all participants who received at least 1 dose of treatment.
Arm/Group | Part 1: Ibrutinib+RICE | Part 1: Ibrutinib+RVICI | Part 2: Ibrutinib+CIT (RICE or RVICI) | Part 2: Chemoimmunotherapy
All-Cause Mortality (participants affected / at risk) | 4/11 | 9/10 | 19/35 | 10/15
Serious Adverse Events (participants affected / at risk) | 10/11 | 9/10 | 25/35 | 11/15
Other Adverse Events (participants affected / at risk) | 11/11 | 10/10 | 35/35 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Ibrutinib+RICE (N=11) | Part 1: Ibrutinib+RVICI (N=10) | Part 2: Ibrutinib+CIT (RICE or RVICI) (N=35) | Part 2: Chemoimmunotherapy (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 3
Febrile Bone Marrow Aplasia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 | 3 | 21 | 6
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 2 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 4
Sinus Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Optic Atrophy (Eye disorders) | 0 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric Ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal Inflammation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Mucosal Inflammation (General disorders) | 0 | 0 | 0 | 1
Multiple Organ Dysfunction Syndrome (General disorders) | 1 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 1
Systemic Inflammatory Response Syndrome (General disorders) | 0 | 0 | 1 | 0
Hepatic Failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Anaphylactic Reaction (Immune system disorders) | 0 | 0 | 1 | 0
Infusion Related Hypersensitivity Reaction (Immune system disorders) | 0 | 0 | 0 | 1
Anorectal Infection (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Capnocytophaga Infection (Infections and infestations) | 0 | 0 | 0 | 1
Corynebacterium Infection (Infections and infestations) | 1 | 0 | 0 | 0
Cryptosporidiosis Infection (Infections and infestations) | 0 | 0 | 1 | 0
Device Related Infection (Infections and infestations) | 0 | 1 | 1 | 1
Escherichia Sepsis (Infections and infestations) | 0 | 0 | 1 | 2
Herpes Zoster (Infections and infestations) | 0 | 1 | 0 | 0
Klebsiella Sepsis (Infections and infestations) | 0 | 1 | 1 | 0
Meningitis (Infections and infestations) | 0 | 1 | 0 | 0
Neutropenic Sepsis (Infections and infestations) | 0 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 3 | 0
Pulmonary Mycosis (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 4 | 5 | 3
Septic Shock (Infections and infestations) | 1 | 0 | 3 | 0
Staphylococcal Infection (Infections and infestations) | 1 | 0 | 0 | 0
Vascular Device Infection (Infections and infestations) | 0 | 0 | 1 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 0 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0 | 0 | 0
Blood Bilirubin Increased (Investigations) | 0 | 1 | 0 | 0
Coagulation Test Abnormal (Investigations) | 0 | 0 | 0 | 1
Neutrophil Count Decreased (Investigations) | 1 | 0 | 1 | 0
Platelet Count Decreased (Investigations) | 1 | 0 | 3 | 1
White Blood Cell Count Decreased (Investigations) | 0 | 0 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Altered State of Consciousness (Nervous system disorders) | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Haemorrhage Intracranial (Nervous system disorders) | 0 | 1 | 0 | 0
Hepatic Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Paraplegia (Nervous system disorders) | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0
Spinal Cord Haematoma (Nervous system disorders) | 0 | 1 | 0 | 0
Subarachnoid Haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Tonic Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0
Toxic Encephalopathy (Nervous system disorders) | 0 | 1 | 1 | 0
Psychotic Disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 1 | 0
Cystitis Haemorrhagic (Renal and urinary disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal Failure (Renal and urinary disorders) | 0 | 1 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Capillary Leak Syndrome (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Ibrutinib+RICE (N=11) | Part 1: Ibrutinib+RVICI (N=10) | Part 2: Ibrutinib+CIT (RICE or RVICI) (N=35) | Part 2: Chemoimmunotherapy (N=15)
Anaemia (Blood and lymphatic system disorders) | 8 | 9 | 29 | 14
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0
Febrile Bone Marrow Aplasia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 5 | 2 | 6 | 1
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 1 | 10 | 3
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Macrocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 6 | 6 | 14 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 8 | 19 | 4
Pericardial Effusion (Cardiac disorders) | 0 | 1 | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 5 | 2
Aplasia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Ear Pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 1 | 0
Eye Pain (Eye disorders) | 0 | 0 | 0 | 1
Eyelid Oedema (Eye disorders) | 1 | 0 | 0 | 0
Eyelid Ptosis (Eye disorders) | 0 | 1 | 0 | 0
Keratitis (Eye disorders) | 0 | 1 | 0 | 0
Pupils Unequal (Eye disorders) | 0 | 0 | 0 | 1
Vision Blurred (Eye disorders) | 1 | 0 | 0 | 0
Xerophthalmia (Eye disorders) | 0 | 1 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 3 | 5 | 12 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 6 | 1
Anal Erythema (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Anal Inflammation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Anal Ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Anorectal Ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Aphthous Ulcer (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Chapped Lips (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 3 | 8 | 3
Dental Caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 6 | 10 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 5 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal Inflammation (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Gastrointestinal Motility Disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gingival Bleeding (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Gingival Oedema (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Mouth Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Mouth Ulceration (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 7 | 5 | 21 | 2
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oesophageal Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 7 | 3
Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 5 | 5 | 25 | 4
Asthenia (General disorders) | 1 | 0 | 2 | 0
Catheter Site Granuloma (General disorders) | 1 | 0 | 0 | 0
Catheter Site Pain (General disorders) | 0 | 0 | 2 | 0
Chest Pain (General disorders) | 0 | 0 | 3 | 2
Chills (General disorders) | 0 | 1 | 0 | 0
Device Related Thrombosis (General disorders) | 0 | 0 | 0 | 1
Face Oedema (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 5 | 0
Generalised Oedema (General disorders) | 1 | 0 | 2 | 1
Hypothermia (General disorders) | 0 | 0 | 0 | 1
Mucosal Inflammation (General disorders) | 2 | 4 | 9 | 3
Mucosal Ulceration (General disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 3 | 3 | 14 | 5
Swelling (General disorders) | 0 | 0 | 0 | 1
Swelling Face (General disorders) | 1 | 0 | 0 | 0
Hepatic Failure (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Drug Hypersensitivity (Immune system disorders) | 0 | 0 | 2 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Hypogammaglobulinaemia (Immune system disorders) | 1 | 1 | 0 | 1
Anal Abscess (Infections and infestations) | 0 | 1 | 0 | 1
Aspergillus Infection (Infections and infestations) | 0 | 0 | 2 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Bk Virus Infection (Infections and infestations) | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0
Device Related Infection (Infections and infestations) | 2 | 0 | 3 | 1
Escherichia Infection (Infections and infestations) | 0 | 0 | 0 | 1
Fungal Infection (Infections and infestations) | 0 | 0 | 0 | 1
Fusarium Infection (Infections and infestations) | 0 | 1 | 0 | 0
Geotrichum Infection (Infections and infestations) | 0 | 1 | 0 | 0
Herpes Zoster (Infections and infestations) | 0 | 2 | 0 | 0
Klebsiella Infection (Infections and infestations) | 1 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 0
Oral Herpes (Infections and infestations) | 0 | 1 | 2 | 1
Pneumonia (Infections and infestations) | 0 | 2 | 1 | 0
Pseudomonal Bacteraemia (Infections and infestations) | 1 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 2
Rhinovirus Infection (Infections and infestations) | 0 | 1 | 2 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0 | 1
Urinary Tract Infection Pseudomonal (Infections and infestations) | 0 | 0 | 0 | 1
Vascular Device Infection (Infections and infestations) | 0 | 1 | 0 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1
Buttock Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Fractured Sacrum (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 | 1 | 4 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 0 | 4 | 0
Transfusion Reaction (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Traumatic Haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 4 | 0 | 7 | 6
Amylase Increased (Investigations) | 0 | 0 | 1 | 1
Antithrombin Iii Decreased (Investigations) | 1 | 1 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 5 | 0 | 6 | 5
Blood Bilirubin Increased (Investigations) | 3 | 1 | 2 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 1 | 0 | 1 | 0
C-Reactive Protein Increased (Investigations) | 1 | 1 | 3 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 2 | 1 | 2 | 0
Haemoglobin Decreased (Investigations) | 1 | 0 | 1 | 0
International Normalised Ratio Increased (Investigations) | 0 | 1 | 1 | 2
Lipase Increased (Investigations) | 0 | 0 | 0 | 1
Lymphocyte Count Decreased (Investigations) | 1 | 0 | 4 | 2
Neutrophil Count Decreased (Investigations) | 1 | 2 | 12 | 9
Pancreatic Enzymes Decreased (Investigations) | 1 | 0 | 0 | 0
Platelet Count Decreased (Investigations) | 5 | 2 | 12 | 8
Staphylococcus Test Positive (Investigations) | 0 | 0 | 0 | 1
Weight Decreased (Investigations) | 0 | 1 | 3 | 0
Weight Increased (Investigations) | 0 | 0 | 1 | 1
White Blood Cell Count Decreased (Investigations) | 1 | 2 | 8 | 6
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 3 | 3 | 0
Fluid Retention (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 5 | 7 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 3 | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 6 | 12 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2 | 6 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 4 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 2 | 5 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 5 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 5 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 7 | 1
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 1
Depressed Level of Consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 2 | 1
Headache (Nervous system disorders) | 1 | 1 | 16 | 3
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 1
Muscle Spasticity (Nervous system disorders) | 0 | 0 | 0 | 1
Myoclonus (Nervous system disorders) | 0 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 1 | 0
Spinal Cord Haematoma (Nervous system disorders) | 0 | 1 | 0 | 0
Toxic Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 0
Confusional State (Psychiatric disorders) | 0 | 0 | 1 | 2
Depression (Psychiatric disorders) | 0 | 1 | 1 | 2
Hallucination (Psychiatric disorders) | 0 | 1 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 4 | 0
Irritability (Psychiatric disorders) | 1 | 0 | 0 | 1
Post-Traumatic Stress Disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 5 | 0
Hypotonic Urinary Bladder (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal Impairment (Renal and urinary disorders) | 0 | 0 | 2 | 1
Renal Tubular Injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Penile Swelling (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 8 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Respiratory Alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 4 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 4 | 2 | 1
Hypotension (Vascular disorders) | 0 | 2 | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will with hold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT02703272/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-04): https://cdn.clinicaltrials.gov/large-docs/72/NCT02703272/SAP_001.pdf